CLINICAL TRIAL: NCT03691714
Title: An Open-label, Phase II Study of Durvalumab (MEDI4736) in Combination With Cetuximab in Previously Treated Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma (HNSCC)
Brief Title: Durvalumab (MEDI4736) With Cetuximab in Previously Treated Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Trisha Wise-Draper (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, Trisha Wise-Draper, Investigator, University of Cincinnati
Organization: University of Cincinnati (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCCI-HN-17-02; EAR-17-12765 (Other Grant/Funding Number: AstraZeneca Pharmaceuticals)
Record Dates: First submitted 2018-09-28; First posted 2018-10-02 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Recurrent Head and Neck Cancer; Head and Neck Cancer; Head and Neck Neoplasms; Metastatic Cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Neoplasm Metastasis | interventions — durvalumab; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Durvalumab and Cetuximab (Experimental): Durvalumab 500mg as a 120-minute intravenous infusion every two weeks. Cetuximab 400mg/m2 IV loading dose followed by weekly Cetuximab 250mg/m2 IV Treatment with Durvalumab continues until progression and Cetuximab may continue as maintenance
  Interventions: Drug: Durvalumab; Drug: Cetuximab

INTERVENTIONS:
Drug: Durvalumab — Two hour infusion
  Other Names: MEDI4736
Drug: Cetuximab — Two hour infusion for loading dose followed by weekly one hour infusion

SUMMARY:
The purpose of this research study is to test the combination of the anti-cancer drugs durvalumab, the study drug, and cetuximab as a treatment for metastatic or recurrent head and neck cancer. Participants will receive both durvalumab and cetuximab.

DETAILED DESCRIPTION:
This research study is designed to see if the study drug, durvalumab, will work better with cetuximab than either medicine alone along with the evaluation of side effects of the drug combination.

ELIGIBILITY:
Inclusion Criteria:

* Body weight > 30 kg
* Histologically or cytologically confirmed recurrent or metastatic HNSCC
* Not considered a candidate for other curative therapy (i.e. surgery/RT)
* Documented progression of disease after receiving platinum based regimen
* ECOG performance status 0-2

Exclusion Criteria:

* Nasopharyngeal and salivary gland tumors
* Prior exposure to both immunotherapy drugs and Cetuximab. Single exposure to either immunotherapy or cetuximab is allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-10-23 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 24 months
  Imaging review using RECIST 1.1

SECONDARY OUTCOMES:
Adverse events | 24 months
  Percentage of adverse events using CTCAE v 5.0
Disease control rate | 6 months
  Combined complete response, partial response, and stable disease
Progression-free survival | 24 months
  Imaging review using RECIST 1.1
Overall survival | 24 months
  Date of on treatment to date of death
Duration of response | 24 months
  Date of initial response to progressive disease

CONTACTS AND LOCATIONS:
Overall Officials: Shuchi Gulati, MD, Principal Investigator — University of Cincinnati
Locations (1):
- UC Health, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No